CLINICAL TRIAL: NCT01103804
Title: A Prospective, Non-interventional Study to Evaluate the Change in Symptoms Scores and Treatment Response After 4 Weeks of Systematic Treatment With PPIs in GERD Patients in Primary Care Setting in Romania, Using the Validated GerdQ Questionnaire.
Brief Title: Non-interventional Study to Evaluate the Change in Symptoms Scores and Treatment Response After 4 Weeks of Proton-Pump Inhibitors (PPI) Treatment
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-GRO-DUM-2009/1
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Gastroesophageal Reflux
Keywords: GerdQ questionnaire
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of the study is to describe the change in GerdQ sum scores, after a 4-week period of systematic treatment with PPIs(using GerdQ questionnaire). The secondary objectives are: to measure the response at the current treatment after a 4-week period of systematic treatment and to identify the percentage of patients which require alterations of their treatment (GerdQ questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Patients known or newly diagnosed with GERD or patients with typical symptoms of GERD- heartburn, regurgitation (in the last case, GerdQ sum score should be ≥8, in the absence of PPI treatment)

Exclusion Criteria:

* Any symptoms at visit 1 suggesting a need for further investigation, judged by the Investigator (alarm symptoms).The alarm symptoms suggesting complicated disease are: dysphagia, odynophagia, bleeding, weight loss without intention or anemia.
* Previous participation in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are patients known/newly diagnosed with GERD or with symptoms suggesting GERD( hearburn, regurgitations) who presented to their family physician(primary care clinic)
Sampling Method: Probability Sample
Enrollment: 952 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
describe the change in GerdQ sum scores, after a 4-week period of systematic treatment with PPIs(GerdQ) | 4 weeks(at V1 and V2)

SECONDARY OUTCOMES:
measure the response at the current treatment after a 4-week period of systematic treatment with PPIs(GerdQ) | 4 weeks(at V1 and V2)
identify the percentage of patients which require alterations of their treatment after a 4-week period of systematic treatment with PPIs(GerdQ) | 4 weeks(at V1 and V2)

CONTACTS AND LOCATIONS:
Overall Officials: CRISTINA TEODORESCU, Study Director — AstraZeneca Pharma SRL Romania
Locations (19):
- Romania (19):
  - Research Site, Arad
  - Research Site, Bacau
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Cluj-Napoca
  - Research Site, Floreşti
  - Research Site, Galati
  - Research Site, Iași
  - Research Site, Piteşti
  - Research Site, Ploieşti
  - Research Site, Rm. Valcea
  - Research Site, Sibiu
  - Research Site, Slatina
  - Research Site, Târgovişte
  - Research Site, Tg. Mures
  - Research Site, Timișoara
  - Research Site, Vanatori(GL)